CLINICAL TRIAL: NCT07248852
Title: Benefits of Guided Movement Using a Maraca of the Arm Opposite to the One Undergoing Venipuncture to Reduce Pain in Children Aged 1-3 Years: a Multicentre Randomized Controlled Trial
Brief Title: Guided Distraction Movement
Acronym: MOVING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP241783; IDRCB 2025-A00034-45 (Other: ANSM)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Venipuncture Pain
Keywords: Active distraction; Venipuncture; Children; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual practice (No Intervention): In this arm, venipuncture will be performed according to usual care. The usual care recommended for young children is as follows:
  * The child is lying down, sitting or in a semi-setting position or in the arms of an adult (parent or health professional).
  * Parents are present if they wish. The child may have his or her cuddly toy.
  * Analgesia is administered using anaesthetic cream and, depending on the child and the department's routine, anaesthetic cream and/or nitroxusmay be added.
  * No distracting objects are used apart from the voice (whispers, unsung words) or reassuring gestures as in usual practice (e. g. caresses, gentle rocking ). No active distraction with a toy or a screen are offered.
  * The child's gestures may be restrained by the professional(s) if necessary, in accordance with the department's policies and current practices. 62 caractères maximum.
  Facultatif si la description de l'intervention (cf. ci-dessous) décrit suffisamment le bras.
- Usual practice and active distraction. (Experimental): Venipuncture will be performed according to the usual care with the addition of active distraction using the maraca.
  Active distraction procedure: The nurse performing the venipuncture called the operator and a professional called the 'accompanying person' (nurse, nursing assistant or childcare assistant usually in charge of looking after or holding the child) sit on either side of the child.
  * At the start of the procedure, the accompanying person places the maraca in the child's hand and shows him/her that it makes a noise 30 seconds before the venipuncture. The accompanying person checks the movement of the child's hand by placing his/her own hand on the child's hand. He/she playfully suggests to the child to wait to make noise with the maraca by counting down 'on 3, we'll make noise'. This countdown allows coordination with the operator.
  * When the operator is ready to perform the venipuncture, the accompanying person invites the child to gently shake the maraca.
  If the venipun
  Interventions: Other: Guided movement

INTERVENTIONS:
Other: Guided movement — Active distraction procedure:
  Venipuncture will be performed according to the usual care with the addition of active distraction using the maraca.
  Active distraction procedure: The nurse performing the venipuncture called the operator and a professional called the 'accompanying person' (nurse, nursing assistant or childcare assistant usually in charge of looking after or holding the child) sit on either side of the child.
  * At the start of the procedure, the accompanying person places the maraca in the child's hand and shows him/her that it makes a noise 30 seconds before the venipuncture. The accompanying person checks the movement of the child's hand by placing his/her own hand on the child's hand. He/she playfully suggests to the child to wait to make noise with the maraca by counting down 'on 3, we'll make noise'. This countdown allows coordination with the operator.
  * When the operator is ready to perform the venipuncture, the accompanying person invites the child to gently sha
  Arms: Usual practice and active distraction.

SUMMARY:
The aim of this research is to evaluate the benefits of using a maraca to guide movement in order to reduce pain during venipuncture for blood sampling or infusion (insertion of a peripheral venous line) in children aged 1 to 3 years.

Pharmacological methods can reduce the pain associated with venipuncture, but they do not address all aspects of pain. Complementary methods have been studied, such as distraction.

According to the literature, interventions in which the child actively participates, with motor action, have been little explored before 3 years of age.

Encouraging children aged 1 to 3 years to perform a movement using a maraca of the arm opposite to the one undergoing venipuncture, in synchronisation with the venipuncture, in addition to current pharmacological methods, would be a simple active intervention.

This distraction method has never been studied. It could reduce pain, withdrawal reactions and also the need for restraint by caregivers, leading to better acceptance of treatment and a higher success rate.

During a multicentre randomized controlled trial conducted in France, the benefits of guided movement using a maraca of the arm opposite to the one undergoing venipuncture synchronised with venipuncture and combined with the usual practice, will be compared with the usual practice alone. 5000 caractères maximum

DETAILED DESCRIPTION:
Pharmacological methods can reduce the pain associated with venipuncture, but they do not address all aspects of pain. Complementary methods have been studied, such as distraction.

According to the literature, distraction interventions are effective in limiting self-reported or reported pain but not behavioural pain. The studies involved children aged 3 years and older who were distracted using passive methods such as reading, listening or watching a video.

On the other hand, in children aged 1 month to 3 years, no passive strategy was found to reduce pain.

Interventions in which the child actively participates, with motor action, have been little explored before 3 years of age.

Encouraging children aged 1 to 3 years to perform a movement using a maraca of the arm opposite to the one undergoing venipuncture, in synchronisation with the venipuncture, in addition to current pharmacological methods, would be a simple active intervention.

This distraction method has never been studied. It could reduce pain, withdrawal reactions and also the need for restraint by caregivers, leading to better acceptance of treatment and a higher success rate.

Based on studies demonstrating the effectiveness of active and multisensory distraction strategies, the hypothesis is based on the fact that voluntary movement, by simultaneously soliciting vision and hearing, captures the child's attention sufficiently to reduce the perception of pain and withdrawal reactions, thereby limiting restraint.

The aim of this study is to evaluate benefits of guided movement using a maraca of the arm opposite to the one undergoing venipuncture synchronised with venipuncture and combined with the usual practice, compared with the usual practice alone in children aged 1 to 3 years.

Two groups will be compared during a multicentre randomized controlled trial conducted in France. One group will receive usual practice with pharmacological analgesia (anaesthetic cream and/or nitroxus). In the other group, the usual practice will be combined with guided movement using a maraca of the arm opposite to the one undergoing venipuncture synchronised with venipuncture.

The evaluation will also include a qualitative analysis of the perceptions of the intervention by the parents and professionals involved.

ELIGIBILITY:
Inclusion Criteria:

* aged 1 to 3 years
* with a venipuncture prescribed within the first 48 hours of hospitalization in general paediatrics or during a consultation

Exclusion Criteria:

* motor disability of upper limbs
* mental disability with neuromotor troubles
* venipuncture or other invasive procedure (lumbar puncture or catheter insertion) within 2 hours prior to inclusion
* more than 5 venipunctures within 48 hours prior to inclusion
* clinical condition requiring emergency venous access

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pain score evaluated from the video recording of the procedure using the FLACC scale, | Day 1
  Pain score evaluated from the video recording of the procedure using the FLACC scale, completed between 2 minutes before the venipuncture and the end of the first venipuncture.
  The assessment will be performed remotely and independently by two expert professionals.

SECONDARY OUTCOMES:
Restraint evaluated using PRIC scale | Day 1
Immobility of the arm undergoing venipuncture evaluated using a numerical scale from 0 to 10 (in the absence of an internationally validated scale). | Day 1
Intensity of the arm withdrawal reaction during venipuncture evaluated using a numerical scale from 0 to 10 (in the absence of an internationally validated scale). | Day 1
Proportion of venipuncture successfully completed at the first attempt. | Day 1
Acceptability of intervention from the child's perspective | Day 1
  Acceptability of intervention from the child's perspective, evaluated by parents and attending professionals (nurses, nursing assistants and childcare assistants ) using a numerical scale from 0 to 10.
Qualitative evaluation conducted through semi-structured interviews with 15 parents (or parental couples) and 15 nurses, nursing assistants or childcare assistants who participated in the intervention. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte LOMBART, Paramedical coordinator, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Direction de la recherche et de l'innovation, Paris, France